CLINICAL TRIAL: NCT01238848
Title: A Randomized Controlled Trial to Evaluate Efficacy of Nebulized Hypertonic Saline vs. Normal Saline in the Treatment of Hospitalized Children With Bronchiolitis
Brief Title: Efficacy of Nebulized Hypertonic Saline in the Treatment of Acute Bronchiolitis
Acronym: Hypertonic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General de Niños Pedro de Elizalde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGNPE-14-2010
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Results first posted 2012-08-17 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2012-07

CONDITIONS: Bronchiolitis
Keywords: Hypertonic; Saline; Bronchiolitis; Efficacy
MeSH Terms: conditions — Bronchiolitis | interventions — Saline Solution, Hypertonic; Saline Solution; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypertonic (Experimental): Nebulized hypertonic saline (sodium chloride 3%) + albuterol
  Interventions: Drug: Hypertonic saline
- Normal (Active Comparator): Normal saline (sodium chloride 0.9%) + albuterol
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Hypertonic saline — 3 cc nebulized hypertonic saline + albuterol 0.25 mg/kg/day, four times a day (QID), 5 days
  Other Names: ClNa 3% (sodium chloride 3%)
  Arms: Hypertonic
Drug: Normal saline — 3 cc nebulized normal saline + albuterol 0.25 mg/kg/day, four times a day (QID), 5 days
  Other Names: ClNa 0.9% (sodium chloride 0.9%)
  Arms: Normal

SUMMARY:
The purpose of this study is to evaluate the efficacy of hypertonic saline vs. normal saline in the treatment of infants hospitalized for bronchiolitis, regarding length of hospital stay, oxygen requirements and clinical outcome.

DETAILED DESCRIPTION:
Despite bronchiolitis is a very frequent disease among infants, there are still controversies regarding its treatment. Hypertonic saline has been proposed as useful treatment in these children, bur information is still controversial.

The aim is to asses that using Nebulized Hypertonic Saline with bronchodilators (albuterol) may reduce the days of hospitalization and improve clinical outcomes in patients with acute bronchiolitis, compared with using Normal Saline with albuterol.

ELIGIBILITY:
Inclusion criteria:

* Infants aged 1 to 24 months, hospitalized for first episode of bronchiolitis, with severity score ≥ 5 points and oxygen saturation ≥ 97%.

Exclusion Criteria:

* Chronic respiratory or cardiovascular disease, respiratory failure.

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria I Espelt, MD, Principal Investigator — Hospital General de Niños Pedro de Elizalde
Locations (1):
- Hospital General de Niños Pedro de Elizalde, Buenos Aires, Buenos Aires F.D., Argentina

REFERENCES:
- [Background] Zhang L, Mendoza-Sassi RA, Wainwright C, Klassen TP. Nebulized hypertonic saline solution for acute bronchiolitis in infants. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD006458. doi: 10.1002/14651858.CD006458.pub2. PMID 18843717
- [Background] Ralston S, Hill V, Martinez M. Nebulized hypertonic saline without adjunctive bronchodilators for children with bronchiolitis. Pediatrics. 2010 Sep;126(3):e520-5. doi: 10.1542/peds.2009-3105. Epub 2010 Aug 16. PMID 20713480
- [Derived] Zhang L, Mendoza-Sassi RA, Wainwright CE, Aregbesola A, Klassen TP. Nebulised hypertonic saline solution for acute bronchiolitis in infants. Cochrane Database Syst Rev. 2023 Apr 4;4(4):CD006458. doi: 10.1002/14651858.CD006458.pub5. PMID 37014057

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypertonic: Hypertonic saline (sodium chloride 0.3%) + albuterol
Period: Overall Study
Arm/Group | Hypertonic | Normal
Started | 50 | 50
Completed | 37 | 45
Not Completed | 13 | 5
Not completed — Physician Decision | 13 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypertonic | Normal | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 50 | 100
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 4.6 (4.1) | 4.2 (2.5) | 4.5 (3.8)
Gender [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 26 | 24 | 50

OUTCOME MEASURES:

1. Secondary Outcome: Length of Oxygen Use
Description: Length of oxygen use (days)
Time Frame: Participants will be followed for the duration of hospitalization, an expected average of 4 days
Measure: Median (Standard Deviation); unit: days
Arm/Group | Hypertonic | Normal
Number analyzed (Participants) | 37 | 45
days | 4 (3.4) | 3.22 (2.3)

2. Primary Outcome: Hospitalization Days
Description: hospitalization days
Time Frame: Participants will be followed for the duration of hospitalization, an expected average of 4 days
Measure: Median (Standard Deviation); unit: days
Arm/Group | Hypertonic | Normal
Number analyzed (Participants) | 37 | 45
days | 5.8 (2.7) | 5.47 (2.1)

ADVERSE EVENTS:
Arm/Group | Hypertonic | Normal
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
The initially estimated sample size was not achieved

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No